CLINICAL TRIAL: NCT03633370
Title: Multifaceted Intervention for Increasing Performance of Cardiopulmonary Resuscitation by Laypersons in Out-of-hospital Cardiac Arrest. A Stepped Wedge Cluster Randomized Controlled Trial
Brief Title: Multifaceted Intervention for Increasing Performance of CPR by Laypersons in Out-of-hospital Cardiac Arrest
Acronym: DISPATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: DISPATCH
Record Dates: First submitted 2018-07-19; First posted 2018-08-16 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Dispatcher; Cardiopulmonary Resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: A Stepped Wedge Cluster Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Usual management of patients according to international guidelines. Protocols of call acceptance, phone advice and sending of emergency services are not modified
- Test Group (Other): Multifaceted intervention
  1. Training using distance learning for medical regulation assistants to recognise cardiac arrest on phone
  2. Activation of the location-software application to send bystanders on cardiac arrest location before the arrival of emergency medical services (EMS)
  3. Motivation feed-back Volunteers will received feed-back regarding CPR initiated before EMS arrival and survival
  Interventions: Other: Multifaceted intervention including 3 components

INTERVENTIONS:
Other: Multifaceted intervention including 3 components — Multifaceted intervention including Dispatcher training to improve cardiac phone recognition, mobile application to send bystanders on cardiac arrest location before first professionals rescuers and motivational support for volunteer bystanders
  Arms: Test Group

SUMMARY:
Cardiac arrest (CA) early recognition is essential in order to rapidly activate emergency services and for bystanders to begin cardiopulmonary resuscitation (CPR).

As soon as a call is received, EMS dispatchers should try to identify CA. This may be difficult, in a context of stress and distress of the person calling. Yet, it is vital for bystanders to initiate CPR. Survival can be multiplied by 2 to 4 if the bystanders initiate a CPR before the arrival of the emergency medical services.

This work aim to assess a multifaceted intervention combining 3 elements to improve the initial phone recognition of CA and raise the number of patients benefiting from CPR before EMS arrival on scene.

The first element is a dispatcher training to the early phone recognition of CA. This training will be based on the concept of active teaching, favouring the interactive work of learners in particular by listening to real dispatch recordings. It will be completed by continuing education with a distance teaching platform including the systematic listening of recorded CA calls.

The second element is based on the deployment of a software aiming to notify CA thanks to mobile phones. This system interfaced to a control software enables to request the participation of CPR-trained volunteers automatically. The volunteers have to be located in the patient's surroundings. The deployment of this mobile application will rely on first-aid volunteers, health personal and any trained volunteers willing to participate. A randomized control study in one city area proved the efficiency of a similar software to improve the proportion of CPR by bystanders.

The third element consists in a motivational feedback. A weekly overview of the management and the outcomes of patients who suffered CA will be broadcast to all the responders and volunteers in the mobile application.

ELIGIBILITY:
Inclusion Criteria:

* All adults with nontraumatic, out-of-hospital cardiac arrest diagnosed during the emergency medical service call
* Cardiac arrest located in urban area

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients under the law
* Patients deprived of liberty by court ruling or administrative ruling
* Traumatic cardiac arrest
* CA occurring under the eyes of a professional emergency services patrol on duty
* Cardiac arrest for which resuscitation seem unjustified (inevitable death, terminally ill irreversible condition, too long duration of cardiac arrest, non-resuscitation personal directive…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2481 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
CPR initiated by bystanders before the arrival of first professionals rescuers | Day 0
  Proportion of patients who's received CPR initiated by bystander before EMS arrival.

SECONDARY OUTCOMES:
Survival at 72h after out-of-hospital cardiac arrest | 72 hours
  survival at 72h
Return of Spontaneous Circulation | Day 0
  Proportion of patients who's recovered a spontaneous circulation after CPR
Survival to hospital admission | Day 0
  Vital status at hospital admission
Survival to hospital discharge | up to 30 days
  Vital status at hospital discharge
Survival at 30 days | 30 days
  Vital status at 30 days
Neurological functional status CPC | up to 30 days
  As measured by Cerebral Performance Category (CPC) at hospital discharge and at 30 days Score less or equal to 2 will be considered as favorable neurological outcome
Neurological functional status mRS | 30 days
  As measured by modified Rankin Scale (mRS) at hospital discharge and at 30 days:
  modified Rankin Scale (mRS): 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead Score less or equal to 3 will be considered as favorable neurological outcome
First recorded rhythm | 30 min
  First recorded cardiac rhythm by EMS

OTHER OUTCOMES:
Bystander's CPR quality | Day 0
  Evaluation of CPR quality performed by bystanders on a 4 points scale. CPR quality will be assessed by first professional rescuers on scene.
Confirmation of cardiac arrest | Days 0
  The dispatcher CA's recognition will be confirmed by EMS on scene
Automated External Defibrillator initiated before EMS arrival | Day 0
  Proportion of patients who's benefit to a automated external defibrillator before the EMS arrivals
CPR initiation by witness without dispatcher Telephone-CPR | Day 0
  Evaluation of the proportion of patients with CPR initiated before EMS arrival without dispatcher Telephone-CPR
CPR initiation by witness with Telephone-CPR | Day 0
  Evaluation of CPR initiated before EMS arrival following Telephone-CPR
CPR initiation by app-activated bystanders | Day 0
  Evaluation of CPR initiated by bystanders, who are activated by the geo-localization application
Proportion of cardiac arrest correctly identified after dispatch | 24 months
  Assessment of the evolution in CA recognition after the e-learning training

CONTACTS AND LOCATIONS:
Overall Officials: Monique Sorentino, Study Director — CHU Grenoble Alpes
Locations (15):
- France (15):
  - SAMU 80 - CHU Amiens Picardie, Amiens
  - SAMU 74 - CH Annecy Genevois, Annecy
  - SAMU 33 - CHU Hôpital Pellegrin, Bordeaux
  - SAMU 01 - CH Fleyriat, Bourg-en-Bresse
  - SAMU 29 - CHRU La Cavale Blanche, Brest
  - SAMU 73 - Centre Hospitalier Métropôle Savoie, Chambéry
  - SAMU 21 - CHU Dijon, Dijon
  - SAMU 38 - CHU Grenoble Alpes, Grenoble
  - Samu 85 - Chd Les Oudairies, La Roche-sur-Yon
  - SAMU 54 - CHU Nancy, Nancy
  - SAMU 44 - Hôtel Dieu, Nantes
  - SAMU 06 - CHU de Nice, Nice
  - SAMU 42 -CHU Saint-Etienne, Saint-Etienne
  - SAMU 31 - CHU Toulouse, Toulouse
  - SAMU 26 - CH de Valence, Valence

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be submitted for publication. IPD will be shared with other researcher.
Supporting Information: Study Protocol, SAP, ICF, CSR